CLINICAL TRIAL: NCT00788957
Title: A Randomized, Phase 1b/2 Trial of AMG 102 or AMG 479 in Combination With Panitumumab Versus Panitumumab Alone in Subject With Wild-Type KRAS Metastatic Colorectal Cancer
Brief Title: Panitumumab Combination Study With Rilotumumab or Ganitumab in Wild-type Kirsten Rat Sarcoma Virus Oncogene Homolog (KRAS) Metastatic Colorectal Cancer (mCRC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NantBioScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060447
Record Dates: First submitted 2008-10-23; First posted 2008-11-11 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Colon Cancer; Colorectal Cancer; Gastrointestinal Cancer; Metastatic Colorectal Cancer; Rectal Cancer
Keywords: panitumumab; vectibix; AMG 102; AMG 479; colon cancer; rectal cancer; colorectal cancer; metastatic colorectal cancer; EGFR inhibitor; IGF inhibitor; c-MET inhibitor
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Rectal Neoplasms | interventions — Panitumumab; ganitumab; rilotumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (6):
- Part 1: Panitumumab + Rilotumumab (Experimental): Participants received panitumumab 6 mg/kg and rilotumumab 10 mg/kg by intravenous infusion once every 2 weeks until progressive disease, intolerability, withdrawal, death or sponsor decision.
  Interventions: Drug: Panitumumab; Drug: Rilotumumab
- Part 2: Panitumumab Alone (Active Comparator): Participants received panitumumab 6 mg/kg and placebo by intravenous infusion once every 2 weeks until progressive disease, intolerability, withdrawal, death or sponsor decision.
  Interventions: Drug: Panitumumab
- Part 2: Panitumumab + Rilotumumab (Experimental): Participants received panitumumab 6 mg/kg and rilotumumab 10 mg/kg by intravenous infusion once every 2 weeks until progressive disease, intolerability, withdrawal, death or sponsor decision.
  Interventions: Drug: Panitumumab; Drug: Rilotumumab; Drug: Placebo
- Part 2: Panitumumab + Ganitumab (Experimental): Participants received panitumumab 6 mg/kg and ganitumab 12 mg/kg by intravenous infusion once every 2 weeks until progressive disease, intolerability, withdrawal, death or sponsor decision.
  Interventions: Drug: Panitumumab; Drug: Ganitumab; Drug: Placebo
- Part 3: Rilotumumab (Experimental): Participants randomized to Panitumumab Alone in Part 2 who had disease progression (radiographic or clinical) or intolerability were re-randomized in Part 3 to receive rilotumumab 10 mg/kg every 2 weeks until disease progression, intolerability, withdrawal, death, or sponsor decision.
  Interventions: Drug: Rilotumumab; Drug: Placebo
- Part 3: Ganitumab (Experimental): Participants randomized to Panitumumab Alone in Part 2 who had disease progression (radiographic or clinical) or intolerability were re-randomized in Part 3 to receive ganitumab 12 mg/kg every 2 weeks until disease progression, intolerability, withdrawal, death, or sponsor decision.
  Interventions: Drug: Ganitumab; Drug: Placebo

INTERVENTIONS:
Drug: Panitumumab — Panitumumab for intravenous infusion
  Other Names: Vectibix®
  Arms: Part 1: Panitumumab + Rilotumumab; Part 2: Panitumumab + Ganitumab; Part 2: Panitumumab + Rilotumumab; Part 2: Panitumumab Alone
Drug: Ganitumab — Ganitumab for intravenous infusion
  Other Names: AMG 479
  Arms: Part 2: Panitumumab + Ganitumab; Part 3: Ganitumab
Drug: Rilotumumab — Rilotumumab for intravenous infusion
  Other Names: AMG 102
  Arms: Part 1: Panitumumab + Rilotumumab; Part 2: Panitumumab + Rilotumumab; Part 3: Rilotumumab
Drug: Placebo — Placebo intravenous infusion
  Arms: Part 2: Panitumumab + Ganitumab; Part 2: Panitumumab + Rilotumumab; Part 3: Ganitumab; Part 3: Rilotumumab

SUMMARY:
This study is a global, multicenter, open-label phase 1b and randomized, double-blinded, 2 part, phase 2 study designed to evaluate the safety and efficacy of rilotumumab or ganitumab in combination with panitumumab versus panitumumab alone in patients with metastatic colorectal cancer whose tumors are wild-type KRAS status.

DETAILED DESCRIPTION:
This study consisted of 3 parts:

Part 1: determination of the tolerable dose of rilotumumab in combination with panitumumab to be administered in Part 2.

Part 2: Comparison of the safety and efficacy of rilotumumab or ganitumab in combination with panitumumab versus that of panitumumab alone. In Part 2, participants were randomized 1:1:1 into 3 cohorts: 6 mg/kg panitumumab plus 10 mg/kg rilotumumab, 6 mg/kg panitumumab plus 12 mg/kg ganitumab, or 6 mg/kg panitumumab and placebo (panitumumab alone cohort). Panitumumab was administered open-label, and rilotumumab and ganitumab were double-blinded.

Part 3: Exploratory evaluation of the safety and efficacy of the rilotumumab and ganitumab monotherapy following treatment with panitumumab in Part 2. In Part 3, eligible participants who terminated panitumumab treatment in the Panitumumab Alone arm of Part 2 due to disease progression or intolerability could be randomized 1:1 into 2 double-blind cohorts: 10 mg/kg rilotumumab or 12 mg/kg ganitumab.

Participants who permanently discontinued all the investigational products completed a safety follow-up visit 30 days and a follow-up visit 60 days after the last dose of investigational product. Participants were followed for radiographic disease progression and survival every 3 months after the 30-day safety follow-up visit for up to 2 years after the last participant was enrolled in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* metastatic adenocarcinoma of the colon or rectum
* wild-type KRAS tumor status
* radiographic evidence of disease progression during or following treatment with irinotecan and/or oxaliplatin containing chemotherapy for mCRC
* measurable disease >/= 20 mm per Response Evaluation Criteria In Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* adequate laboratory values

Exclusion Criteria:

* history of central nervous system (CNS) metastases
* history of another primary cancer, unless:
* curatively resected non-melanomatous skin cancer
* curatively treated cervical carcinoma in situ
* other primary solid tumor treated with curative intent and no known active disease present for >/= 5 years
* prior treatment with an anti-epithelial growth factor receptor (EGFR), hepatocyte growth factor receptor (HGFR, c-MET), and/or insulin-like growth factor receptor (IGFR) inhibitor
* prior treatment with AMG 102 or AMG 479
* prior treatment with chemotherapy or radiotherapy </= 21 days
* prior treatment with targeted therapy </= 30 days
* known allergy or hypersensitivity to panitumumab, AMG 102, or AMG 479
* history of interstitial lung disease
* clinically significant cardiovascular disease </= 1 year
* active inflammatory bowel disease
* known human immunodeficiency virus (HIV), hepatitis C, or hepatitis B infection
* any co-morbid disease or condition that could increase the risk of toxicity
* serious or non-healing wound </= 35 days
* any uncontrolled concurrent illness or history of any medical condition that could interfere with the interpretation of the study results
* major surgical procedure </= 35 days or minor surgical procedure </= 14 days
* other investigational procedures or drugs </= 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2008-10-27 (Actual); Primary Completion 2010-07-23 (Actual); Study Completion 2010-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Van Cutsem E, Eng C, Nowara E, Swieboda-Sadlej A, Tebbutt NC, Mitchell E, Davidenko I, Stephenson J, Elez E, Prenen H, Deng H, Tang R, McCaffery I, Oliner KS, Chen L, Gansert J, Loh E, Smethurst D, Tabernero J. Randomized phase Ib/II trial of rilotumumab or ganitumab with panitumumab versus panitumumab alone in patients with wild-type KRAS metastatic colorectal cancer. Clin Cancer Res. 2014 Aug 15;20(16):4240-50. doi: 10.1158/1078-0432.CCR-13-2752. Epub 2014 Jun 11. PMID 24919569
- [Derived] Peeters M, Kafatos G, Taylor A, Gastanaga VM, Oliner KS, Hechmati G, Terwey JH, van Krieken JH. Prevalence of RAS mutations and individual variation patterns among patients with metastatic colorectal cancer: A pooled analysis of randomised controlled trials. Eur J Cancer. 2015 Sep;51(13):1704-13. doi: 10.1016/j.ejca.2015.05.017. Epub 2015 Jun 3. PMID 26049686
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24919569/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 27 October 2008; last patient enrolled 05 February 2010. In Part 1, participants with wild-type KRAS metastatic colorectal cancer received open-label rilotumumab and panitumumab to identify a tolerable dose of rilotumumab for Part 2 of the study. Participants enrolled in Part 1 were not eligible for randomization in Part 2.
Pre-assignment Details: In Part 2 participants were randomized in a 1:1:1 ratio to the 3 double-blinded treatment arms. In Part 3, participants randomized to Panitumumab Alone in Part 2 and with disease progression or intolerability were re-randomized 1:1 into 2 double-blind groups.
  Clinically significant laboratory findings were considered adverse events, so the protocol endpoint "Incidence of all AEs and clinical laboratory abnormalities" was not analyzed separately but was included in the AE data
Period: Part 1
Arm/Group | Part 1: Panitumumab + Rilotumumab | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab | Part 3: Rilotumumab | Part 3: Ganitumab
Started | 11 | 0 | 0 | 0 | 0 | 0
Completed | 2 (Completed the safety follow-up visit) | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Panitumumab + Rilotumumab | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab | Part 3: Rilotumumab | Part 3: Ganitumab
Started | 0 | 48 | 48 | 46 | 0 | 0
Completed | 0 | 6 (Completed the safety follow-up visit at the end of the study) | 4 (Completed the safety follow-up visit) | 5 (Completed the safety follow-up visit) | 0 | 0
Not Completed | 0 | 42 | 44 | 41 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 9 | 5 | 3 | 0 | 0
Not completed — Death | 0 | 32 | 35 | 37 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0 | 0
Not completed — On-study at time of data cut-off | 0 | 1 | 1 | 1 | 0 | 0
Period: Part 3
Arm/Group | Part 1: Panitumumab + Rilotumumab | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab | Part 3: Rilotumumab | Part 3: Ganitumab
Started | 0 | 0 | 0 | 0 | 13 | 11
Completed | 0 | 0 | 0 | 0 | 4 (Completed the safety follow-up visit) | 1 (Completed the safety follow-up visit)
Not Completed | 0 | 0 | 0 | 0 | 9 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 8 | 8
Not completed — On-study at time of data cut-off | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set, including participants who received at least one dose of respective investigational product in the corresponding parts of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Panitumumab + Rilotumumab | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab | Part 3: Rilotumumab | Part 3: Ganitumab | Total
Number analyzed (Participants) | 11 | 48 | 48 | 46 | 13 | 11 | 177
Age, Continuous [Mean (Standard Deviation); unit: years]
  Part 1 Participants | 56.5 (13.8) | NA (NA) | NA (NA) | NA (NA) | NA (NA) | NA (NA) | 56.5 (13.8)
  Part 2 Participants | NA (NA) | 55.0 (12.5) | 62.1 (7.5) | 62.0 (9.7) | NA (NA) | NA (NA) | 59.7 (10.6)
  Part 3 Participants | NA (NA) | NA (NA) | NA (NA) | NA (NA) | 54.8 (13.9) | 52.0 (11.3) | 53.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 20 | 19 | 21 | 3 | 6 | 75
  Male | 5 | 28 | 29 | 25 | 10 | 5 | 102
Race/Ethnicity, Customized [Number; unit: participants] — Hispanic/Latino was collected as Race Category.
  participants
    White or Caucasian | 11 | 45 | 47 | 45 | 13 | 10 | 171
    Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 2
    Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Other | 0 | 1 | 0 | 0 | 0 | 1 | 2
Subjects With Wild-Type KRAS Metastatic Colorectal Cancer [Count of Participants; unit: Participants] | 11 | 48 | 48 | 46 | 13 | 11 | 177

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicities (DLT)
Description: A DLT is defined as any grade 3 or 4 rilotumumab-related or combination (panitumumab and rilotumumab)-related adverse event or laboratory abnormality that is deemed clinically significant by the investigator
Time Frame: 7 weeks
Population: The first 6 DLT evaluable participants, including participants who received at least 2 doses of panitumumab and rilotumumab as scheduled (ie, Week 1 and 3) and have a minimum 28 days follow-up for safety or, have received at least 1 dose of panitumumab and rilotumumab and had a DLT within the first 28 days on study.
Measure: Number; unit: participants
Arm/Group | Part 1: Panitumumab + Rilotumumab
Number analyzed (Participants) | 6
participants | 0

2. Primary Outcome: Part 2: Percentage of Participants With an Objective Response
Description: An objective response is defined as a confirmed complete (CR) or partial response (PR) no less than 4 weeks after the criteria for response are first met, determined by the investigator considering the radiologic response of all existing target and non-target lesions, evidence of new lesions, and cytology evaluation (as appropriate) according to the Modified-Response Evaluation Criteria In Solid Tumors (RECIST) v1.0 criteria: CR: Disappearance of all target and non-target and no new lesions. PR: At least a 30% decrease in the size of target lesions with no increase in non-target lesions, or, the disappearance of all target lesions and persistence of one or more non-target lesion(s) not qualifying for either CR or progressive disease. Participants without a post-baseline assessment were considered non-responders. Tumor assessments up to the initiation of another anti-tumor therapy including the Part 3 treatment, if applicable, were used.
Time Frame: From the date of first dose until the data cut-off date of 23 July 2010. Median follow-up time was 30 weeks.
Population: Efficacy analysis set (enrolled participants who received at least one dose of respective investigational product in the corresponding parts of the study) with measurable baseline disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 48 | 48 | 46
percentage of participants | 21 [10.5 to 35.0] | 31 [18.7 to 46.3] | 22 [10.9 to 36.4]

3. Secondary Outcome: Duration of Response - Part 2
Description: Time from the confirmed objective response to disease progression per the modified RECIST v1.0 criteria.
Time Frame: From the date of first dose until the data cut-off date of 23 July 2010. Median follow-up time was 30 weeks.
Population: Only subjects with confirmed response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 10 | 15 | 10
Months | 3.7 [3.6 to NA] — Not estimable as number of responding subjects and number with events was too small to calculate upper confidence interval. | 5.1 [3.7 to 5.6] | 3.7 [3.6 to 5.8]

4. Secondary Outcome: Time to Response - Part 2
Description: Time from the first dose of investigational product to the date of first confirmed objective response. Calculated only for subject with a confirmed objective response
Time Frame: From the date of first dose until the data cut-off date of 23 July 2010. Median follow-up time was 30 weeks.
Population: Only subjects with confirmed response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 10 | 15 | 10
Months | 1.8 [1.6 to 2.5] | 1.6 [1.6 to 1.7] | 1.7 [1.6 to 1.7]

5. Secondary Outcome: Disease Control Rate - Part 2
Description: The incidence of confirmed objective response or stable disease. Stable disease cannot be established prior to study day 49 (calculated from the date of first dose of investigational product), ie, the earliest protocol scheduled tumor assessment
Time Frame: From the date of first dose until the data cut-off date of 23 July 2010. Median follow-up time was 30 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 48 | 48 | 46
percentage of participants | 56 [41 to 71] | 71 [56 to 83] | 61 [45 to 75]

6. Secondary Outcome: Progression-free Survival (PFS) - Part 2
Description: Time from the first dose of investigational product to the date of disease progression per the modified RECIST v1.0 criteria or death
Time Frame: From the date of first dose until the data cut-off date of 23 July 2010. Median follow-up time was 30 weeks.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 48 | 48 | 46
Months | 3.7 [2.5 to 5.3] | 5.2 [3.6 to 5.4] | 5.3 [2.7 to 5.7]

7. Secondary Outcome: On-treatment Progression-free Survival (PFS) - Part 2
Description: Time from the first dose of investigational product to the date of disease progression per the modified RECIST v1.0 criteria or death during the treatment period (from the first to last dose of investigational product). Radiographic progression within 28 days since last dose of study therapy (last component of combination therapy) up to the initiation of another anti-tumor therapy, including the Part 3 treatment, if applicable, or death within 28 days since last dose of study therapy.
Time Frame: From the date of first dose until the data cut-off date of 23 July 2010. Up to 56 weeks.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 48 | 48 | 46
Months | 3.8 [2.5 to 5.3] | 5.3 [3.6 to 5.4] | 5.3 [2.7 to 5.7]

8. Secondary Outcome: Overall Survival - Part 2
Description: The interval in months from the first dose of investigational product to the date of death.
Time Frame: From the date of first dose until the data cut-off date of 23 July 2010. Median follow-up time was 30 weeks.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 48 | 48 | 46
Months | NA [8.6 to NA] — Median and upper CIs are not estimable due to small number of subjects with events in time period. | NA [9.6 to NA] — Median and upper CIs are not estimable due to small number of subjects with events in time period. | NA [7.1 to NA] — Median and upper CIs are not estimable due to small number of subjects with events in time period.

9. Secondary Outcome: Cmin, Cmax of Panitumumab
Description: Cmin = minimum drug concentration during a dosing interval; Cmax = maximum observed drug concentration during a dosing interval
Time Frame: 14 days
Population: PK population
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Part 1: Panitumumab + Rilotumumab
Number analyzed (Participants) | 6
μg/mL
  Cmin | 42.5 [32.2 to 105]
  Cmax | 223 [166 to 276]

10. Secondary Outcome: Cmin, Cmax, for Rilotumumab
Description: as for outcome 9
Time Frame: 14 days
Population: PK population
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Part 1: Panitumumab + Rilotumumab
Number analyzed (Participants) | 6
μg/mL
  Cmin | 120 [86.7 to 171]
  Cmax | 306 [264 to 488]

11. Secondary Outcome: Cmin for Panitumumab - Part 2
Description: Cmin = minimum drug concentration during a dosing interval
Time Frame: Up to 23 weeks
Population: PK population Measure of dispersion is %CV
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 43 | 42 | 44
μg/mL
  Week 3 | 19.8 (80.3) | 22.8 (73.5) | 17.2 (56.5)
  Week 5 | 34.8 (58.9) | 37.9 (52.5) | 29.8 (55.7)
  Week 7 | 39.9 (62.2) | 45.2 (50.4) | 37.4 (54.5)
  Week 13 | 63.5 (43.0) | 63.4 (45.2) | 51.4 (63.1)
  Week 23 | 82.1 (28.2) | 62.1 (44.3) | 54.8 (53.8)

12. Secondary Outcome: Cmax for Panitumumab - Part 2
Description: Cmax = maximum observed drug concentration during a dosing interval
Time Frame: Up to 23 weeks
Population: PK population Measure of dispersion is %CV
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 43 | 42 | 44
μg/mL
  Week 1 | 114 (27.7) | 124 (26.4) | 118 (34.7)
  Week 3 | 149 (31.4) | 154 (29.0) | 139 (24.4)
  Week 5 | 165 (30.1) | 172 (32.3) | 150 (26.5)
  Week 7 | 166 (30.8) | 180 (29.6) | 167 (23.9)
  Week 13 | 201 (26.7) | 199 (25.7) | 192 (31.2)
  Week 23 | 196 (24.5) | 207 (24.9) | 187 (22.3)

13. Secondary Outcome: Cmin for Rilotumumab - Part 2
Description: Cmin = minimum drug concentration during a dosing interval
Time Frame: Up to 23 weeks
Population: PK population Measure of dispersion is %CV
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 2: Panitumumab + Rilotumumab
Number analyzed (Participants) | 43
μg/mL
  Week 3 | 70.1 (41.2)
  Week 5 | 119 (31.8)
  Week 7 | 143 (27.5)
  Week 13 | 186 (40.7)
  Week 23 | 181 (36.3)

14. Secondary Outcome: Cmax for Rilotumumab - Part 2
Description: Cmax = maximum observed drug concentration during a dosing interval
Time Frame: Up to 23 weeks
Population: PK population Measure of dispersion is %CV
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Part 2: Panitumumab + Rilotumumab
Number analyzed (Participants) | 43
μg/ml
  Week 1 | 239 (29.3)
  Week 3 | 316 (28.4)
  Week 5 | 357 (25.0)
  Week 7 | 397 (24.8)
  Week 13 | 453 (23.7)
  Week 23 | 421 (26.0)

15. Secondary Outcome: Cmin for Ganitumab - Part 2
Description: Cmin = minimum drug concentration during a dosing interval
Time Frame: Up to 23 weeks
Population: PK population Measure of dispersion is %CV
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 42
μg/ml
  Week 3 | 19.8 (51.6)
  Week 5 | 24.4 (55.2)
  Week 7 | 28.9 (54.2)
  Week 13 | 38.8 (61.6)
  Week 23 | 39.7 (58.8)

16. Secondary Outcome: Cmax for Ganitumab - Part 2
Description: Cmax = maximum observed drug concentration during a dosing interval
Time Frame: Up to 23 weeks
Population: PK population Measure of dispersion is %CV
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 42
μg/mL
  Week 1 | 218 (30.0)
  Week 3 | 240 (25.3)
  Week 5 | 244 (29.3)
  Week 7 | 279 (35.5)
  Week 13 | 274 (28.1)
  Week 23 | 276 (22.8)

17. Secondary Outcome: Total Anti-Panitumumab Antibody Incidence - Part 2
Description: Ratio of the number of subjects with at least one positive antibody result at baseline (or at any post-baseline or long-term follow-up time point) to the number of subjects with at least one immunoassay results at baseline (or at any post-baseline or long term follow-up time point). Measured by either Biacore or ELISA.
Time Frame: First dose of any study drug and before 120 days of last dose of study drugs; up to 1 year, eight months
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 48 | 48 | 46
percentage of participants | 6.3 | 18.8 | 17.4

18. Secondary Outcome: Total Anti-AMG 102 Antibody Incidence - Part 2
Description: Ratio of the number of subjects with at least one positive antibody result at baseline (or at any post-baseline or long-term follow-up time point) to the number of subjects with at least one immunoassay results at baseline (or at any post-baseline or long term follow-up time point). Measured by MSD.
Time Frame: First dose of any study drug and before 120 days of last dose of study drugs, up to 1 year, eight months.
Population: Only subjects having AMG-102 treatment in part 2 were measured for antibody incidence.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Panitumumab + Rilotumumab
Number analyzed (Participants) | 48
percentage of participants | 6.3

19. Secondary Outcome: Total Anti-AMG 479 Antibody Incidence - Part 2
Description: as for outcome 18
Time Frame: First dose of any study drug and before 120 days of last dose of study drugs, up to 1 year, eight months.
Population: Only subjects having AMG-479 treatment in part 2 were measured for antibody incidence.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Panitumumab + Ganitumab
Number analyzed (Participants) | 46
percentage of participants | 17.4

20. Secondary Outcome: AUC for Rilotumumab
Description: AUC = area under the drug concentration-time curve during a dosing interval
Time Frame: 14 Days
Population: PK population
Measure: Median (Full Range); unit: day•μg/mL
Arm/Group | Part 1: Panitumumab + Rilotumumab
Number analyzed (Participants) | 6
day•μg/mL | 2300 [2020 to 3540]

21. Secondary Outcome: AUC for Panitumumab
Description: AUC = area under the drug concentration-time curve during a dosing interval
Time Frame: 14 Days
Population: PK Population
Measure: Median (Full Range); unit: day•μg/mL
Arm/Group | Part 1: Panitumumab + Rilotumumab
Number analyzed (Participants) | 6
day•μg/mL | 1200 [987 to 1890]

ADVERSE EVENTS:
Time Frame: All non-serious AEs that occurred after initiation of investigational product through 30 days after the last dose of investigational product or the 30-day safety follow-up visit, whichever was later, up to 56 weeks. All serious AEs that occurred after the subject signed the informed consent form through 30 days after the last dose of investigational product or the 30-day safety follow-up visit, whichever was later, up to 56 weeks.
Arm/Group | Part 1: Panitumumab + Rilotumumab | Part 2: Panitumumab Alone | Part 2: Panitumumab + Rilotumumab | Part 2: Panitumumab + Ganitumab | Part 3: Rilotumumab | Part 3: Ganitumab
All-Cause Mortality (participants affected / at risk) | 8/11 | 32/48 | 35/48 | 37/46 | 8/13 | 8/11
Serious Adverse Events (participants affected / at risk) | 5/11 | 11/48 | 9/48 | 9/46 | 6/13 | 2/11
Other Adverse Events (participants affected / at risk) | 11/11 | 42/48 | 47/48 | 44/46 | 11/13 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Panitumumab + Rilotumumab (N=11) | Part 2: Panitumumab Alone (N=48) | Part 2: Panitumumab + Rilotumumab (N=48) | Part 2: Panitumumab + Ganitumab (N=46) | Part 3: Rilotumumab (N=13) | Part 3: Ganitumab (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Eastern cooperative oncology group performance status worsened (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercreatininaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Panitumumab + Rilotumumab (N=11) | Part 2: Panitumumab Alone (N=48) | Part 2: Panitumumab + Rilotumumab (N=48) | Part 2: Panitumumab + Ganitumab (N=46) | Part 3: Rilotumumab (N=13) | Part 3: Ganitumab (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 7 | 2 | 1 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 3 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 6 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 5 | 3 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 5 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 11 | 5 | 6 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 7 | 11 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 8 | 4 | 3 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 4 | 6 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 7 | 3 | 5 | 1 | 0
Asthenia (General disorders) | 3 | 7 | 4 | 6 | 0 | 5
Chills (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Fatigue (General disorders) | 4 | 10 | 4 | 8 | 1 | 3
Infusion related reaction (General disorders) | 2 | 0 | 0 | 4 | 0 | 0
Mucosal inflammation (General disorders) | 3 | 3 | 6 | 5 | 0 | 0
Oedema peripheral (General disorders) | 2 | 6 | 9 | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 4 | 2 | 2 | 1 | 2
Paronychia (Infections and infestations) | 4 | 7 | 15 | 9 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 5 | 1 | 0
Weight increased (Investigations) | 0 | 3 | 1 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 8 | 10 | 9 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 6 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 1 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5 | 6 | 4 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 10 | 13 | 19 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 0 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 4 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 6 | 0 | 1 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 3 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 4 | 0 | 2 | 1 | 0
Depression (Psychiatric disorders) | 0 | 4 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 5 | 5 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 3 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 7 | 2 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 5 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 16 | 17 | 12 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 7 | 11 | 10 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3 | 4 | 5 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 12 | 10 | 13 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 25 | 28 | 22 | 3 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 8 | 7 | 12 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 2 | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 2 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 1 | 2 | 2 | 1 | 1
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 1 | 2 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 2 | 2 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Genital tract inflammation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Koilonychia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Part 3 of the study did not reach the accrual goal. Only 24 out of the 42 planned subjects received treatment in Part 3 of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT00788957/Prot_SAP_000.pdf